CLINICAL TRIAL: NCT06418945
Title: Porphyromonas Gingivalis Elimination From Oral Improves Esophageal Cancer Patients Survival After Radical Operation
Brief Title: Clinical Study on the Effect of Removal of Porphyromonas Gingivalis on Prognosis of Esophageal Cancer After Radical Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGESCC001
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Evaluate the DFS of Patients With Esophageal Cancer Who Underwent Radical Operation After Regular Removal of Porphyromonas Gingivalis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1:pg（-） (No Intervention): The routine follow-up review after radical resection of esophageal cancer was performed according to the schedule requirements
- Arm 2:pg（+） (Experimental): Dental cleaning combined with gum tape treatment every three months until disease progression/recurrence/death or intolerable adverse reactions occur.
  Interventions: Combination Product: Tinidazole oral microneedle patch
- Arm 3:pg（+） (No Intervention): The routine follow-up review after radical resection of esophageal cancer was performed according to the schedule requirements

INTERVENTIONS:
Combination Product: Tinidazole oral microneedle patch — Ultrasonic teeth cleaning: After gargling with compound chlorhexidine gargle or 3% hydrogen peroxide gargle for 1 minute, the teeth were cleaned by ultrasonic wave. After the teeth were cleaned, the wound was rinsed with 3% hydrogen peroxide to stop bleeding. Immediately after the ultrasonic cleaning, two pieces of tinidazole oral composite microneedle patch were applied to the upper and lower gums close to the inside of the first molar, especially on the tooth loss or damage, and the mouth was kept closed for 15 minutes. After the microneedle was fully degraded, the room could be left.
  Other Names: Ultrasonic tooth cleaning
  Arms: Arm 2:pg（+）

SUMMARY:
Esophagectomy is an important means of radical treatment of esophageal cancer, but due to local recurrence and metastasis, the 5-year survival rate of patients with esophageal cancer is only 20-30%. Studies have reported that about 50% of patients relapse within 1 year after surgery, and the short-term recurrence rate is high. Therefore, reducing the recurrence rate of esophageal cancer after operation is an important way to improve its prognosis. Porphyromonas gingivalis infection in ESCC tissues was significantly higher than that in paracancer tissues, and was significantly positively correlated with cancer cell differentiation, lymph node metastasis, TNM stage, and shortened survival of ESCC patients. In summary, porphyromonas gingivalis plays an important role in postoperative recurrence of esophageal cancer. Elimination of porphyromonas gingivalis can significantly reduce the recurrence rate of esophageal cancer after operation. Tinidazole is a class of nitroimidazole drugs. It has been pointed out that the pharmacological mechanism of Tinidazole is to inhibit the DNA synthesis of pathogenic bacteria, so as to eliminate bacteria in periodontal tissues and inhibit local inflammation. Based on this, we designed and fabricated a novel oral microneedle patch loaded with tinidazole. Tinidazole oral microneedle patch can effectively remove porphyromonas gingivalis and promote the repair of gingival tissue. In this study, based on the combination of mechanical removal and antibacterial treatment, a combination of ultrasonic dental cleaning and tinidazole oral composite microneedle patch was designed to completely remove porphyromonas gingivalis in oral cavity, and to evaluate the effect of removal of porphyromonas gingivalis in oral cavity on the prognosis of esophageal cancer after radical surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85 years old
2. Histologically confirmed esophageal cancer
3. Patients undergoing radical resection for esophageal cancer who do not require or are not eligible for radiotherapy，T1-T4N0-3M0
4. ECOG：0～1
5. Expected survival ≥12 weeks
6. Radical surgery was performed within 28 days and met R0 criteria
7. The patient did not receive neoadjuvant radiotherapy/neoadjuvant concurrent chemoradiotherapy before surgery and no longer received adjuvant radiotherapy/adjuvant chemoradiotherapy
8. If the major organs function normally, the following criteria are met: HB≥90g/L；b.ANC≥1.5×109/L；c.PLT ≥80×109/L；ALB≥30g/L；b.ALT和AST≤2.5ULN
9. Women of reproductive age should agree to use contraceptives (such as Iuds, contraceptives, or condoms) during the study period and for 6 months after the study ends; Have a negative serum or urine pregnancy test within 7 days prior to study enrollment and must be a non-lactating patient; Men should consent to patients who must use contraception during the study period and for 6 months after the end of the study period
10. The subjects voluntarily joined the study, signed informed consent, had good compliance, and cooperated with follow-up

Exclusion Criteria:

1. Does not meet the above inclusion criteria
2. Patients with distant visceral metastases
3. Patients requiring adjuvant radiotherapy after neoadjuvant radiotherapy or radical surgery
4. Allergic to tinidazole or metabolic disorder
5. Patients in need of warfarin anticoagulation and those unable to abstain from alcohol
6. Patients who do not tolerate ultrasonic dental cleaning
7. Pregnant or lactating women
8. Patients with other malignancies within 5 years (except cured basal cell carcinoma of the skin and cervical carcinoma in situ)
9. Patients with a history of psychotropic substance abuse who are unable to abstain or have mental disorders
10. Patients who have participated in clinical trials of other drugs within four weeks
11. Patients with concomitant diseases that, in the investigator's judgment, seriously endanger patient safety or interfere with the patient's completion of the study
12. Patients with recurrent mouth ulcers or other oral diseases that affect the oral flora
13. Patients with chronic infectious diseases or autoimmune diseases requiring prolonged or repeated use of antimicrobials or glucocorticoids
14. The researchers did not consider it suitable for inclusion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS | 5 years
  Disease-free survival

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol